CLINICAL TRIAL: NCT06124599
Title: Identification of Prodromal Clinical Signs of Menstrual Staphylococcal Toxic Shock
Brief Title: Prodromes of Menstrual Staphylococcal Toxic Shock
Acronym: IPro-CTSm
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1008
Record Dates: First submitted 2023-10-26; First posted 2023-11-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Toxic Shock Syndrome Staphylococcal
Keywords: Menstrual toxic shock; Staphylococcus aureus; prodromes
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women who have developed menstrual staphylococcal toxic shock: Clinical diagnosis of staphylococcal toxic shock syndrome: "confirmed" or "probable" according to CDC criteria :
  The 5 CDC clinical criteria for Staphylococcal Toxic Shock are:
  * a fever above 39°C,
  * arterial hypotension,
  * generalized scarlatiniform erythroderma
  * intense desquamation of the palms or soles of the feet 7 to 14 days later,
  * and systemic manifestations (at least three):
    * Digestive: vomiting, diarrhea
    * Muscular: myalgias, increased serum creatine phospho-kinase
    * Vaginal, oropharyngeal and conjunctival mucosal hyperemia
    * Renal: hyperuricemia, hypercreatininemia, leukocyturia without urinary infection,
    * Hepatic: increased transaminases
    * Hematological: thrombocytopenia (< 100,000 platelets/mm3)
    * Neurological: excluding episodes of fever or hypotension such as disorientation or altered consciousness.
  If 4 criteria are met, the case is considered probable, and if 5 criteria are met, confirmed.
  Interventions: Other: Identification of symptoms of menstrual staphylococcal toxic shock in last three menstrual period
- Control healthy women: Women over 13 years of age, menstruating and using internal sanitary protection with No history of menstrual toxic shock for controls
  Interventions: Other: Identification of symptoms of menstrual in control patient in the last three menstrual period

INTERVENTIONS:
Other: Identification of symptoms of menstrual staphylococcal toxic shock in last three menstrual period — questionnaire including : fever felt or measured; chills; malaise or feeling of malaise (dizziness when standing up); unusual fatigue; headache; confusion, disorientation; nausea; vomiting; diarrhea; abdominal pain; muscle pain, aches; sore throat or pain when swallowing; red tongue or mouth ulceration; skin rashes (redness, patches...); other
  Groups: Women who have developed menstrual staphylococcal toxic shock
Other: Identification of symptoms of menstrual in control patient in the last three menstrual period — questionnaire including : fever felt or measured; chills; malaise or feeling of malaise (dizziness when standing up); unusual fatigue; headache; confusion, disorientation; nausea; vomiting; diarrhea; abdominal pain; muscle pain, aches; sore throat or pain when swallowing; red tongue or mouth ulceration; skin rashes (redness, patches...); other...
  Groups: Control healthy women

SUMMARY:
Menstrual staphylococcal toxic shock is a rare but severe disease, requiring intensive care in over 80% of cases. Menstrual staphylococcal toxic shock develops during the peri-menstrual period, in healthy young women colonized by a vaginal strain of Staphylococcus aureus secreting the Toxic shock syndrome toxin 1 (TSST-1) and not immune to it, in a favorable environment, i.e. wearing intravaginal menstrual protection (tampon, menstrual cup).

The rarity of the syndrome, its polymorphous clinical presentation and the absence of a totally specific biological examination make menstrual staphylococcal toxic shock a difficult pathology to diagnose. The reference clinical criteria correspond to the advanced picture of multivisceral failure, making it possible to classify cases a posteriori, but contribute to diagnostic delay and lack sensitivity.

Patient accounts suggest the presence of symptoms in the days preceding the development of toxic shock, and also during previous menstrual cycles.

The identification of prodromal symptoms could enable earlier management of menstrual staphylococcal toxic shock by removal of intra-vaginal sanitary protection, the main risk factor, before the disease becomes permanently established and requires intensive care.

ELIGIBILITY:
Inclusion Criteria :

+Case inclusion criteria:

* Women between 13 and 30 years old inclusive
* Clinical diagnosis of staphylococcal toxic shock syndrome: "confirmed" or "probable" according to Center Disease Control (CDC) criteria:

The 5 CDC clinical criteria for menstrual Staphylococcal Toxic Shock are:

* a fever above 39°C,
* arterial hypotension,
* generalized scarlatiniform erythroderma
* intense peeling of the palms or soles of the feet 7 to 14 days later,
* and systemic manifestations (at least three):

  * Digestive: vomiting, diarrhea
  * Muscular: myalgia, increase in serum creatine phosphokinase
  * Hyperemia of the vaginal, oropharyngeal and conjunctival mucous membranes
  * Renal: hyperuricemia, hypercreatininemia, leukocyturia without urinary infection,
  * Hepatic: increase in transaminases
  * Hematological: thrombocytopenia (< 100,000 platelets/mm3)
  * Neurological: apart from episodes of fever or hypotension such as disorientation or altered consciousness.

In the presence of 4 criteria, the case is considered probable and 5 criteria as confirmed case.

* Detection of S. aureus strain carrying Toxic shock syndrome toxin-1 (TSST1) on vaginal samples.
* Onset of symptoms ≤ 72 hours before the start of menstruation and ≥ 72 hours after the end of menstruation.
* Use during the last 3 cycles of vaginal protection: tampon or menstrual cup.

  +Control inclusion criteria:
* Women between 13 and 30 years old inclusive
* Presence of menstruation
* Use of intimate periodic protection, tampon or menstrual cup, during the last 3 periods
* No history of toxic menstrual shock

Exclusion Criteria:

* Non-menstruating women
* Women protected by law
* Women (or relatives) who oppose the study

Ages: 13 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who develop menstrual toxic shock will be identified by reporting their disease to the national staphylococcal reference center by their physician
Sampling Method: Non-Probability Sample
Enrollment: 316 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Women with No history of menstrual toxic shock for controls | in the week following the last menstrual period
  A single collection of information through a questionnaire delivered to the last menstrual period
Patient with Menstrual Staphylococcal Toxic Shock (STC) | in the week following onset Staphylococcal Toxic Shock
  A single collection of information through a questionnaire delivered as close as possible to the occurrence of the STC

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Nord Croix Rousse, Lyon, France